CLINICAL TRIAL: NCT03847233
Title: A Prospective, Multicenter, Single-arm Clinical Trial of Jetstream Atherectomy System for the Treatment of Japanese Patients With Symptomatic Occlusive Atherosclerotic Lesions in the Superficial Femoral and/ or Proximal Popliteal Arteries
Brief Title: Safety and Effectiveness of Jetstream Atherectomy System (J-SUPREME II)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S2450
Record Dates: First submitted 2019-02-18; First posted 2019-02-20 (Actual); Results first posted 2020-12-28 (Actual); Last update posted 2021-08-16 (Actual); Status verified 2021-08

CONDITIONS: Peripheral Arterial Disease
Keywords: Superficial Femoral Artery; Proximal Popliteal Artery; Endovascular therapy; Atherectomy
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Jetstream Atherectomy System (Experimental)
  Interventions: Device: Jetstream Atherectomy System

INTERVENTIONS:
Device: Jetstream Atherectomy System — A rotating, aspirating, expandable catheter system for active removal of atherosclerotic debris and thrombus in the SFA and/or PPA

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of the Jetstream Atherectomy System for the treatment of Japanese patients with symptomatic occlusive atherosclerotic lesions in native superficial femoral artery (SFA) and/ or proximal popliteal arteries (PPA).

DETAILED DESCRIPTION:
A prospective, multicenter, single-arm trial evaluating the safety and efficacy of the Jetstream Atherectomy System in the treatment of symptomatic occlusive atherosclerotic lesions ≤150 mm in length located in the femoropopliteal arteries in subjects with symptoms classified as Rutherford categories 2-4.

ELIGIBILITY:
Inclusion Criteria:

* Chronic, symptomatic lower limb ischemia defined as Rutherford categories 2-4
* Stenotic, restenotic or occlusive lesion(s) located in the native SFA and/or PPA of which meet the following criteria:
* Severely calcified lesions with degree of stenosis ≥70%
* Vessel diameter ≥3.0 mm and ≤6.0 mm
* Total lesion length (or series of lesions) ≤150 mm

Exclusion Criteria:

* Target lesion/vessel with in-stent restenosis
* History of major amputation in the target limb
* Subject has a history of coagulopathy or hypercoagulable bleeding disorder
* Subject with untreatable hemorrhagic disease or platelet count <80,000mm3 or >600,000mm3 as baseline assessment.
* History of myocardial infarction, or stroke/cerebrovascular accident (CVA) within 6 months prior to study enrollment
* Unstable angina pectoris at the time of the enrollment
* Septicemia at the time of enrollment
* Presence of other hemodynamically significant outflow lesions in the target limb requiring a planned surgical intervention or endovascular procedure within 30 days after the index procedure
* Presence of aneurysm in the target vessel
* Acute ischemia and/or acute thrombosis of the SFA/PPA prior to the index procedure
* Perforated vessel as evidenced by extravasation of contrast media prior to the index procedure

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2019-03-19 (Actual); Primary Completion 2019-11-08 (Actual); Study Completion 2020-05-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kazushi Urasawa, MD, PhD, Principal Investigator — Tokeidai Memorial Hospital
Locations (5):
- Japan (5):
  - Tokyo Bay Urayasu Ichikawa Medical Center, Urayasu, Chiba
  - Kokura Memorial Hospital, Kokura, Fukuoka
  - Tokeidai Memorial Hospital, Sapporo, Hokkaido
  - Kansai Rosai Hospital, Amagasaki, Hyōgo
  - Kasukabe Chuo General Hospital, Kasukabe, Saitama

IPD SHARING:
Plan to Share IPD: No
The confidentiality of records/data obtained in the trial will remain anonymous for analysis and publication.
  The information and data, obtained from the trial is used without personal identification.

RESULTS

PARTICIPANT FLOW:
Period: Index Procedure
Arm/Group | Jetstream Atherectomy System
Started | 31
Completed | 31
Not Completed | 0
Period: 6 Month After Index Procedure
Arm/Group | Jetstream Atherectomy System
Started | 31
Completed | 30
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Jetstream Atherectomy System
Number analyzed (Participants) | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.5 (7.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 24
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Japanese | 31
Region of Enrollment [Number; unit: participants]
  Japan | 31
History of renal insufficiency (Hemodialysis) [Count of Participants; unit: Participants] | 7

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Lesion Success
Time Frame: during procedure
Population: Based on the per-protocol analysis set
Measure: Count of Participants; unit: Participants
Groups:
- Jetstream Atherectomy System on the PP Analysis Set: Jetstream Atherectomy System: A rotating, aspirating, expandable catheter system for active removal of atherosclerotic debris and thrombus in the SFA and/or PPA
Arm/Group | Jetstream Atherectomy System on the PP Analysis Set
Number analyzed (Participants) | 28
Participants | 22

2. Other Pre Specified Outcome: Assisted Primary Patency
Time Frame: 1 month and 6 months
Population: One subject did not complete the 6-months follow-up.
Measure: Count of Participants; unit: Participants
Groups:
- Jetstream Atherectomy System on the ITT Analysis Set: Jetstream Atherectomy System: A rotating, aspirating, expandable catheter system for active removal of atherosclerotic debris and thrombus in the SFA and/or PPA
Arm/Group | Jetstream Atherectomy System on the ITT Analysis Set
Number analyzed (Participants) | 31
Participants
  1 month | 31
  6 months: number analyzed (Participants) | 30
  6 months | 29

3. Other Pre Specified Outcome: Primary Patency
Time Frame: 1 month and 6 months
Population: One subject did not complete the 6-months follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Jetstream Atherectomy System on the ITT Analysis Set
Number analyzed (Participants) | 31
Participants
  1 month | 31
  6 months: number analyzed (Participants) | 30
  6 months | 29

4. Other Pre Specified Outcome: Rate of Hemodynamic Improvement
Description: Rate of Hemodynamic Improvement as assessed by changes in Ankle-Brachial Index (ABI) as compared to baseline at 1 month and 6 months
Time Frame: 1 month and 6 months
Population: One subject did not complete the 6-months follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Jetstream Atherectomy System on the ITT Analysis Set
Number analyzed (Participants) | 31
Participants
  1 month | 23
  6 months: number analyzed (Participants) | 30
  6 months | 22

5. Other Pre Specified Outcome: Rate of Primary Sustained Clinical Improvement
Time Frame: 1 month and 6 months
Population: One subject did not complete the 6-months follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Jetstream Atherectomy System on the ITT Analysis Set
Number analyzed (Participants) | 31
Participants
  1 month | 30
  6 months: number analyzed (Participants) | 30
  6 months | 30

6. Other Pre Specified Outcome: Distribution of Rutherford Class
Description: Distribution of Rutherford Class at 1 month and 6 months
Time Frame: 1 month and 6 months
Population: One subject did not complete the 6-months follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Jetstream Atherectomy System on the ITT Analysis Set
Number analyzed (Participants) | 31
Participants
  1 month: Category 0 (Asymptomatic) | 25
  1 month: Category 1 (Mild claudication) | 4
  1 month: Category 2 (Moderate claudication) | 2
  6 months: number analyzed (Participants) | 30
  6 months: Category 0 (Asymptomatic) | 24
  6 months: Category 1 (Mild claudication) | 5
  6 months: Category 2 (Moderate claudication) | 1

7. Other Pre Specified Outcome: Adverse Event Rates
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Jetstream Atherectomy System on the ITT Analysis Set
Number analyzed (Participants) | 31
Participants | 16

8. Other Pre Specified Outcome: Clinically-driven Target Vessel Revascularization (TVR) Rate
Time Frame: 1 month and 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Jetstream Atherectomy System on the ITT Analysis Set
Number analyzed (Participants) | 31
Participants
  1 month | 0
  6 months | 0

9. Other Pre Specified Outcome: Clinically-driven TLR Rate
Time Frame: 1 month and 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Jetstream Atherectomy System on the ITT Analysis Set
Number analyzed (Participants) | 31
Participants
  1 month | 0
  6 months | 0

10. Other Pre Specified Outcome: Major Adverse Event (MAE) Rate
Description: All-cause death through 1 month, and/or target limb major amputation and/or Target Lesion Revascularization (TLR) through 6 months
Time Frame: 1 month and 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Jetstream Atherectomy System on the ITT Analysis Set
Number analyzed (Participants) | 31
Participants
  1 month | 0
  6 months | 0

11. Other Pre Specified Outcome: Reduction in Lesion Stenosis
Description: Change in the percent stenosis prior to treatment with Jetstream and the percent stenosis following treatment with Jetstream (Reduction in Lesion Stenosis=Pre-Jetstream percent stenosis - Post-Jetstream percent stenosis).
Time Frame: Assessed at prior to treatment with Jetstream and after treatment with Jetstream
Measure: Mean (Standard Deviation); unit: percent diameter stenosis
Arm/Group | Jetstream Atherectomy System on the ITT Analysis Set
Number analyzed (Participants) | 31
percent diameter stenosis | 34.6 (16.0)

12. Other Pre Specified Outcome: Number of Patients With Distal Emboli Requiring Additional Treatment
Time Frame: during procedure or within 24 hours post-index procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Jetstream Atherectomy System on the ITT Analysis Set
Number analyzed (Participants) | 31
Participants | 2

13. Other Pre Specified Outcome: Number of Patients With Procedural Success
Time Frame: during procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Jetstream Atherectomy System on the ITT Analysis Set
Number analyzed (Participants) | 31
Participants | 31

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Jetstream Atherectomy System on the ITT Analysis Set
All-Cause Mortality (participants affected / at risk) | 0/31
Serious Adverse Events (participants affected / at risk) | 3/31
Other Adverse Events (participants affected / at risk) | 3/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Jetstream Atherectomy System on the ITT Analysis Set (N=31)
Angina pectoris (Cardiac disorders) | 1
Coronary artery thrombosis (Cardiac disorders) | 1
Pneumonia (Infections and infestations) | 1
Fracture (Injury, poisoning and procedural complications) | 1
Hepatic cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Peripheral artery occlusion (Vascular disorders) | 1 — Left brachial Shunt occlusion
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Jetstream Atherectomy System on the ITT Analysis Set (N=31)
Peripheral embolism (Vascular disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The restriction depends on the conditions on the Clinical Study Agreement at each site. The PI must notify the sponsor about the publication and receive the approval from the sponsor prior to any results/data relavant to the J-SUPREME II trial to be in public.

DOCUMENTS (2):
  • Study Protocol (2019-07-04): https://cdn.clinicaltrials.gov/large-docs/33/NCT03847233/Prot_002.pdf
  • Statistical Analysis Plan (2019-12-13): https://cdn.clinicaltrials.gov/large-docs/33/NCT03847233/SAP_003.pdf